CLINICAL TRIAL: NCT03565471
Title: Atrial Septal Defect - Exercise Capacity and Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-21
Record Dates: First submitted 2018-06-18; First posted 2018-06-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2019-06

CONDITIONS: Atrial Septal Defect; Pulmonary Hypertension
Keywords: Atrial Septal Defect; Exercise Capacity; Pulmonary Hypertension; Heart Rate Variability; Congenital Heart Disease
MeSH Terms: conditions — Heart Septal Defects, Atrial; Hypertension, Pulmonary; Heart Defects, Congenital | interventions — Echocardiography; Exercise Test; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD patients with surgical closure: Patients diagnosed with an ASD who have had a surgical closure of the defect more than 3 years ago.
  Echocardiography, right side catheterization, exercise testing and Holter monitoring are performed on all participants.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right side catheterization; Diagnostic Test: Exercise test; Diagnostic Test: Holter monitor
- ASD patients with transcatheter closure: Patients diagnosed with an ASD who have had a transcatheter closure of the defect more than 3 years ago.
  Echocardiography, right side catheterization, exercise testing and Holter monitoring are performed on all participants.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right side catheterization; Diagnostic Test: Exercise test; Diagnostic Test: Holter monitor
- Controls: Controls who do not have any cardiac or pulmonary diagnoses nor use prescription drugs that may affect the cardiopulmonary function.
  Echocardiography, right side catheterization, exercise testing and Holter monitoring are performed on all participants.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right side catheterization; Diagnostic Test: Exercise test; Diagnostic Test: Holter monitor

INTERVENTIONS:
Diagnostic Test: Echocardiography — Standard echocardiography.
Diagnostic Test: Right side catheterization — Right side catheterization with the purpose of measuring pulmonary vascular pressures and blood saturation.
Diagnostic Test: Exercise test — Exercise test on a supine bicycle with gradual increase in work load while wearing a mask that measures ventilation, oxygen uptake, carbon dioxide release and respiratory exchange rate.
Diagnostic Test: Holter monitor — Holter monitor worn for 2 whole days registering heart rate.

SUMMARY:
The purpose of the study is to compare exercise capacity, cardiac contractility, pulmonary vascular pressures and heart rate variability between patients with an atrial septal defect and healthy controls.

DETAILED DESCRIPTION:
1. Background Patients born with atrial septal defect (ASD) in the heart, have long been assumed healthy after closure of their defect. However, recent studies show, that despite closure of the ASD the risks of arrhythmia, stroke and pneumonia are increased. It is also shown that ASD patients die earlier than the background population and the cause of death is most often cardiac. The reason for this higher mortality and morbidity is unknown and the scope of this thesis.
2. Aim To determine if closed (both surgical and transcatheter) ASD patients have reduced exercise capacity, impaired right and left ventricular function, increased pressure in the pulmonary system, and reduced heart rate variability when compared with healthy controls. The investigators will also examine if method of closure is of importance.
3. Hypothesis

   Primary endpoint:

   The shunting effect alters the hemodynamic in the ASD heart resulting in lower cardiopulmonary exercise capacity when compared with healthy controls.

   Secondary endpoints:

   The shunting effect alters the hemodynamic in the ASD heart when compared with healthy controls resulting in
   * Impaired force frequency relationship with a reduction in contractility at optimal heart rate.
   * Increased pulmonary arterial pressure.
   * Twice as many ASD patients with decreased heart rate variability.

   Surgical closure is thought to have a higher impact on the ventricular function than catheter closure resulting in
   * Lower contractility in the surgically closed patients as compared to the catheter closure as evaluated by force frequency.
   * Twice as many surgically closed patients with decreased heart rate variability compared to catheter closed patients.
4. Materials and methods

   4.1) Power calculation The number of participants needed in the project is calculated based on the exercise capacity test, which is the primary endpoint.

   The normal exercise test result is 48 ml O2/kg/min with a standard deviation of 7 ml O2/kg/min. With an expected difference between groups and healthy controls of 15% and a power of 85%, the number of patients needed in each group is 18. Possible drop-outs are taken into account and therefore 20 participants will be included in each ASD group, they will each be matched one to one with controls, resulting in a total of 80 project participants.

   The secondary endpoints are of a more explorative character, why 20 ASD patients in each group is assumed to be sufficient.

   4.2) Exercise capacity, force frequency relationship and pulmonary hypertension 4.2.1) The exercise capacity test is conducted on a semi-supine bicycle, while the patients wears a mask measuring the ventilation, oxygen uptake, carbon dioxide release and respiratory exchange rate. Patients pedal until maximal exhaustion, which should be obtained after 8-12 minutes.

   4.2.2) During exercise testing, the force frequency relationship is examined using echocardiography.

   4.2.3) A Swan-Ganz catheter is used to measure right-sided hemodynamic pressures and blood saturation.

   4.3) Heart rate variability Electrocardiographic (ECG) activity and heart rate variability will be monitored using a 2-channel Holter monitor. The data will be analyzed with the Pathfinder analysis software.
5. Statistical analysis Results for each group will be expressed as means standard deviation or median range or 95% confidence intervals. One way analysis of variance (ANOVA), paired t-tests and regression analyses will be performed. Analyses will be adjusted for age and sex. The issue of multiple testing/multiple comparisons may arise and only relevant comparisons and analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above.
* Informed consent to participate.
* Patients: Diagnosed with an atrial septal defect. More than 3 years have passed since closure of the atrial septal defect.
* Controls: No history of heart or lung disease.

Exclusion Criteria:

* Lung disease.
* Ischemic heart disease.
* Diabetes.
* Hypertension.
* Valve pathology.
* Patients: Concomitant heart disease
* Controls: Usage of prescription drugs interfering with the cardiopulmonary function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The ASD patients will be identified through the Danish National Patient Registry (DNPR) and enrolled. The controls will be identified from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (ml O2/kg/min) | 8-12 minutes
  using exercise testing
Peak exercise minute ventilation (ml/min) | 8-12 minutes
  using exercise testing
Peak heart rate (beats/min) | 8-12 minutes
  using exercise testing
Maximal workload (W/kg) | 8-12 minutes
  using exercise testing

SECONDARY OUTCOMES:
Tricuspid annular peak systolic velocity (mm) | 8-12 minutes
  using echocardiography
Return gradient at the tricuspid valve (mmHg) | 8-12 minutes
  using echocardiography
Cardiac output (L/min) | 8-12 minutes
  using right sided catheterization
Cardiac index (L/min) | 8-12 minutes
  using right sided catheterization, derived measure adjusted for body surface area
Central venous pressure (mmHg) | 8-12 minutes
  using right sided catheterization
Pulmonary artery wedge pressure (mmHg) | 8-12 minutes
  using right sided catheterization
Pulmonary artery pressure (mmHg) | 8-12 minutes
  using right sided catheterization
Mixed venous oxygen saturation (%) | 8-12 minutes
  using right sided catheterization
Heart rate variability | 48 hours
  using Holter monitoring
Heart rate, minimum, maximum and mean (beats/min) | 48 hours
  using Holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Zarmiga Karunanithi, MD, Principal Investigator — University of Aarhus
Locations (1):
- Dept. of Cardiothoracic & Vascular Surgery, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Karunanithi Z, Andersen MJ, Mellemkjaer S, Alstrup M, Waziri F, Skibsted Clemmensen T, Elisabeth Hjortdal V, Hvitfeldt Poulsen S. Elevated Left and Right Atrial Pressures Long-Term After Atrial Septal Defect Correction: An Invasive Exercise Hemodynamic Study. J Am Heart Assoc. 2021 Jul 20;10(14):e020692. doi: 10.1161/JAHA.120.020692. Epub 2021 Jul 14. PMID 34259012
- [Derived] Alstrup M, Karunanithi Z, Maagaard MO, Poulsen SH, Hjortdal VE. Sympathovagal imbalance decades after atrial septal defect repair: a long-term follow-up study. Eur J Cardiothorac Surg. 2021 Dec 27;61(1):83-89. doi: 10.1093/ejcts/ezab235. PMID 34015096